CLINICAL TRIAL: NCT04861545
Title: Effect of Soy Protein and Its Food Sources on Established Therapeutic Blood Lipid Targets: A Systematic Review and Meta-analysis of Randomized Controlled Trials
Brief Title: Meta-analyses of Soy Protein and Its Food Sources for Cholesterol Reduction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: John Sievenpiper (Other)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Associate Professor, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: Dupont - Soy protein/ISP
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Dyslipidemias; Cardiovascular Risk Factor; Dysglycemia
Keywords: Cardiovascular disease; Coronary heart disease; LDL-Cholesterol; HDL-Cholesterol; Triglycerides; Apolipoprotein B; Soy protein; Isolated soy protein; Meta-analysis; Randomized controlled trial
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Soy — Isolated soy protein food sources are foods that include isolated soy protein in different forms and matrix (e.g. soy beverage and meat analogue).
  Non-isolated soy protein food sources of soy protein are foods made with soy (e.g. Tofu, tempeh, edamame).
  Other Names: Isolated soy protein food sources; Non-Isolated soy protein food sources of soy protein

SUMMARY:
Although soy protein has approved health claims in Canada and the US, and is recognized by major cardiovascular clinical practice guidelines for the reduction of cholesterol and risk of coronary heart disease (CHD), these claims are based almost exclusively on evidence from foods containing isolated soy protein (ISP). The role of other non-ISP food sources of soy protein (e.g Tofu, tempeh, edamame) in these effects is unclear. The role of food form and matrix (e.g soy beverage versus meat analogue) on the effects of ISP is also unclear. As national dietary guidelines and clinical practice guidelines for nutrition therapy shift from a focus on single nutrients to a focus on foods and dietary patterns, it is important to understand whether non-ISP food sources of soy protein and ISP food sources with different food matrices produce the same reductions in LDL-cholesterol and CHD risk. To strengthen the evidence-base for health claims and guidelines development, the investigators will conduct a systematic review and meta-analysis of randomized controlled trials of the effect of ISP and non-ISP food sources of soy protein on stablished lipid targets in individuals with and without dyslipidemia.

DETAILED DESCRIPTION:
RATIONALE. Although soy protein has approved health claims in Canada and the US and is recognized by major cardiovascular clinical practice guidelines for the reduction of cholesterol and risk of coronary heart disease (CHD), these claims are based almost exclusively on evidence from foods containing isolated soy protein (ISP). The role of other non-ISP food sources of soy protein (e.g Tofu, tempeh, edamame) in these effects is unclear. The role of food form and matrix (e.g soy beverage versus meat analogue) on the effects of ISP is also unclear. As national dietary guidelines and clinical practice guidelines for nutrition therapy shift from a focus on single nutrients to a focus on foods and dietary patterns, it is important to understand whether non-ISP food sources of soy protein and ISP food sources with different food matrices produce the same reductions in LDL-cholesterol and CHD risk. The investigators are not aware of any systematic reviews and meta-analyses of randomized controlled trials that have addressed this important question.

OBJECTIVES. To conduct a systematic review of the effect of soy protein with prespecified analyses by food source on established lipid targets in individuals with and without dyslipidemia and assess the certainty of the evidence using the Grading of Recommendations Assessment Development and Evaluation (GRADE) system. A sub-objective is to conduct a targeted systematic review and meta-analysis of the effect of exclusively ISP on established lipid targets in individuals with and without dyslipidemia for use in the development of Health Claims submissions in Australia and New Zealand by co-investigator, Dr. Alan Barclay.

DESIGN. The systematic review and meta-analyses will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting items for Systematic Reviews and Meta-Analyses (PRISMA).

DATA SOURCES. Medline, Embase, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by manual searches of references of included studies.

STUDY SELECTION. Randomized controlled trials of ≥3-weeks (based on the FDA minimum follow-up requirement) assessing the effect of soy protein food sources compared with a suitable non-soy-containing control on lipids will be included.

DATA EXTRACTION. Two or more investigators will independently extract relevant data. Authors will be contacted for additional information and any missing data will be computed/imputed using standard formulae.

RISK OF BIAS. Two or more investigators will independently assess risk of bias using the Cochrane Risk of Bias Tool.

OUTCOMES. The primary outcome will be LDL-C and secondary outcomes will be other established therapeutic lipid targets: HDL-C, TG, non-HDL-D and apo B.

DATA SYNTHESIS. Data will be pooled using the Generic Inverse Variance method with prespecified analyses by food source. Separate pooled analyses will be conducted for ISP to meet the subobjective of assessing the effect of ISP. Random effects models will be used with paired analyses applied to crossover designs. Heterogeneity will be assessed (Cochran Q statistic) and quantified (I2 statistic). Sources of heterogeneity will be explored by sensitivity analyses and a priori subgroup analyses (dose, comparator, follow-up, baseline levels, design, body weight change, saturated fat intake, and risk of bias). Meta-regression will assess the significance of subgroup analyses. Linear and nonlinear dose-response analyses will be assessed by generalized least squares trend (GLST) estimation models and spline curve modelling (MKSPLINE procedure), respectively. Publication bias will be assessed by inspection of funnel plots and the Egger and Begg tests. Adjustment for evidence of funnel plot asymmetry or small study effects will be conducted by the Duval and Tweedie trim-and-fill method.

GRADE ASSESSMENT. To assess the certainty of the evidence, the investigators will use the GRADE system, an evidence-based grading system adopted by >100 organizations (http://www.gradeworkinggroup.org/). It grades the evidence as high, moderate, low or very low quality based on the study design and a series of downgrades (risk of bias, imprecision, inconsistency, indirectness, publication bias) and upgrades (large magnitude of the effect, dose-response gradient, and attenuation by confounding). The investigators will follow the GRADE handbook (https://gdt.gradepro.org/app/handbook/handbook.html) and use the GRADEpro GDT (gradepro.org) software.

KNOWLEDGE TRANSLATION PLAN. The investigators will follow the Ottawa model of Research for knowledge translation. The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact journals. Target audiences will include public health and clinical communities with an interest in nutrition and cardiovascular disease. Feedback will be incorporated and used to improve public health messages and key areas for future research will be defined. The PIs will network among opinion leaders to increase awareness and participate directly in the development of future guidelines.

SIGNIFICANCE. The proposed project will reinforce the role of the all soy protein food sources (not just ISP-containing food sources) for cholesterol and CHD risk reduction, strengthening the evidence-base for health claims and guidelines development in the U.S., Canada, Europe, and beyond and improving health outcomes, by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Randomized controlled trials
* Soy protein (Isolated soy protein and non-isolated soy protein) intervention
* Non-soy protein containing comparator
* Intervention duration ≥ 3 weeks
* Data for at least 1 outcome

Exclusion Criteria:

* Non-human studies
* Observational studies
* Acute single-bolus feeding studies
* Participants <18 years of age
* Interventions of soy derivatives or extracts (i.e. soy oil, sterols, etc)
* No quantification of soy protein in intervention
* Multimodal interventions
* Lack of a suitable comparator (i.e. a comparator arm that contains soy protein)
* Intervention duration < 3 weeks
* No viable outcome data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with and without dyslipidemia
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
1. Blood lipids - LDL-Cholesterol (LDL-C) | ≥ 3 weeks
  LDL-C mean difference and 95%CIs in mmol/L

SECONDARY OUTCOMES:
2. Blood lipids - HDL-Cholesterol (HDL-C) | ≥ 3 weeks
  HDL-C mean difference and 95% CI in mmol/L
3. Blood lipids - Triglycerides (TG) | ≥ 3 weeks
  TG mean difference and 95% CI in mmol/L
4. Blood lipids - Non-HDL-Cholesterol (Non-HDL-C) | ≥ 3 weeks
  Non-HDL-C mean difference and 95% CI in mmol/L
5. Blood lipids - Apolipoprotein B (Apo B) | ≥ 3 weeks
  Apo B mean difference and 95% CI in g/L

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD,PhD,FRCPC, Principal Investigator — University of Toronto; David JA Jenkins, MD,DSc,FRSC, Principal Investigator — University of Toronto; Cyril WC Kendall, PhD, Study Chair — University of Toronto; Alan Barclay, PhD, Study Chair — University of Sydney
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Micheal's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no individual data collected. However, data from all included studies will be published in the manuscript and supplementary material